CLINICAL TRIAL: NCT06242379
Title: Safety and Efficacy Evaluation of Intravitreal Injection of GMP-compliant Bone Marrow Mesenchymal Stem Cell-derived Small Extracellular Vesicles in Patients With Retinitis Pigmentosa
Brief Title: Safety and Efficacy of Stem Cell Small Extracellular Vesicles in Patients With Retinitis Pigmentosa
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R016534006
Record Dates: First submitted 2024-01-12; First posted 2024-02-05 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis pigmentosa; small extracellular vesicles
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bone marrow-mesenchymal stem cell-derived small extracellular vesicles (Experimental): Single intravitreal injection of Good Manufacturing Practice (GMP) compliant bone marrow (BM)-mesenchymal stem cell (MSC)-derived small extracellular vesicles (sEVs) (50 μg) for single eye
  Interventions: Biological: GMP compliant-BM-MSC derived sEVs

INTERVENTIONS:
Biological: GMP compliant-BM-MSC derived sEVs — The procedure will be performed under topical anesthesia (0.5% tetracaine hydrochloride ophthalmic solution). The intravitreal injection will be performed by the retina specialist. Topical antiseptic (5% povidone iodine solution) will be applied on the periorbital and ocular surface. Eyelid speculum will be inserted to expose the injection area. It will include an intravitreal injection at the superotemporal quadrant (right eye) and superonasal quadrant (left eye), 3.5 to 4 mm posterior to the limbus. A 30-gauge needle will be used to deliver a 0.05 to 0.1 ml sEV suspension into the vitreous cavity. Indirect ophthalmoscopy will be performed immediately after the procedure to ensure no occlusion of the central retinal artery. The eye will be rinsed thoroughly by normal saline to wash out remaining antiseptic. The total duration for an intravitreal injection will be approximately 30 minutes.

SUMMARY:
The aim of this clinical trials is to evaluate the safety and efficacy of intravitreal injection of GMP-compliant BM-MSC-derived sEVs in patients with retinitis pigmentosa.

DETAILED DESCRIPTION:
Inherited retinal disease (IRD) is one of the leading causes of blindness in adolescents and adults, affecting 1 in 2,000 to 3,000 people globally. Recently, advances arose in the use of stem cells as treatment modalities for inherited retinal diseases, including retinitis pigmentosa (RP).

The first step, production and characterization of GMP-compliant bone marrow mesenchymal stem cell (BM-MSC)-derived small extracellular vesicles (sEVs) has been performed according to the ethical clearance by the institutional review board of the Faculty of Medicine Siriraj Hospital Mahidol University (approval number Certificate of Approval (COA) no. Si 57112022, protocol number 44312565 (1RB1), dated August 8, 2022). In a prior study, the investigators have conducted a phase I clinical trial to assess the safety of intravitreal autologous MSC injection in 14 patients with advanced-stage RP. After follow-up periods ranging from 1.5 to 7 years, the investigators found that this intervention appeared to be safe and potentially effective. Nevertheless, several mild and one severe adverse event were observed, although all were manageable. Beside the primary outcome, safety of the MSCs, the investigators found statistically significant improvements in the best corrected visual acuity (BCVA) compared to baseline, although they returned to the baseline at 12 months. To minimize the unwanted effects and still maintain the benefit of the MSCs, the cell-free approach using the extracellular vesicles of MSCs is of interest.

On the current study, the investigators would like to evaluate the safety and efficacy of intravitreal injection of GMP-compliant BM-MSC-derived sEVs in patients with retinitis pigmentosa.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Clinically diagnosed with RP by experienced ophthalmologists or having documented mutations in the genes responsible for RP
* Central visual field in the better eye less than or equal to 20 degrees
* Best corrected visual acuity (BCVA) in the worse eye 6/18 (logMAR 0.48) to 6/120 (logMAR 1.3) by Snellen visual acuity chart
* Electroretinogram in the worse eye nonrecordable or the amplitudes were less than 25% of normal
* Willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Intolerance and/or contraindication to local anesthesia and other substances used during the procedure
* Pregnant or lactating woman
* Having blood-borne infections, i.e. Human immunodeficiency virus (HIV), hepatitis B or C, Human T-lymphotropic viruses (HTLV)
* Having any other significant ocular or non-ocular disease/disorder which may either put the subjects at risk because of participation in the study, or may influence the results of the study, or the subjects ability to participate in the study. This includes

  1. Inherited or acquired bleeding disorders, including the use of anticoagulant medications that cannot be stopped prior the procedure
  2. Autoimmune diseases, i.e., systemic lupus erythematosus, multiple sclerosis, fibromyalgia, Guillain-Barre syndrome
  3. Severe/uncontrolled chronic/metabolic diseases, e.g., diabetes mellitus, cardiovascular disease, chronic kidney disease, transient ischemic attack (TIA)/stroke
* Unable to complete the full course of the study or failed to return for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 1 year
  To evaluate the safety of the intervention. The evaluations include the intraocular pressure in mmHg, cell value in number of cells in 0.5 cubic millimeter and flare value in photons per millisecond, anterior segment examination using slit lamp biomicroscopy, fundus evaluation using fundus photography, retinal assessment, and subjective complaints of study participants.
Ophthalmological parameters | 1 year
  To observe the efficacy of the intervention. The evaluations comprise the best corrected visual acuity (BCVA) in the Logarithm of the Minimum Angle of Resolution (LogMAR) score. The value "0" indicates "no loss", that is visual acuity equal to the reference standard (1.0, 20/20). Visual acuity better tans 1.0 (20/20) is represented by negative LogMAR values. LogMAR 1.0 is equivalent to 20/200. Blindness is defined as a best-corrected visual acuity worse than 1.3 LogMAR.
Ophthalmological parameters | 1 year
  contrast sensitivity test using the Stereo Optical Functional Vision Analyzer (FVA) to measure contrast sensitivity by generating a contrast sensitivity function curve that portrays sensitivity on the Y-axis and spatial frequency on the X-axis.
Ophthalmological parameters | 1 year
  sweep visual evoked potential in Snellen unit
Ophthalmological parameters | 1 year
  kinetic visual field test in degree field of vision at four quadrants (superior, nasal, inferior, temporal)
Ophthalmological parameters | 1 year
  optic disc and cup volume in cubic millimeter
Ophthalmological parameters | 1 year
  retinal nerve fiber layer thickness in micron
Ophthalmological parameters | 1 year
  electrophysiology (electroretinography in microvolt, visual evoked potential in millisecond and microvolt, multifocal electroretinography in signal strength response)
Ophthalmological parameters | 1 year
  optical coherence tomography of the macula in micron
Ophthalmological parameters | 1 year
  optical coherence tomography angiography in percent of vessel flow density
Ophthalmological parameters | 1 year
  foveal avascular zone in square millimeter
Ophthalmological parameters | 1 year
  macular thickness in micron

CONTACTS AND LOCATIONS:
Overall Officials: Laongsri Atchaneeyasakul, Professor, Principal Investigator — Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Need a consensus from colleagues; Personal reasons

REFERENCES:
- [Background] Cremers FPM, Boon CJF, Bujakowska K, Zeitz C. Special Issue Introduction: Inherited Retinal Disease: Novel Candidate Genes, Genotype-Phenotype Correlations, and Inheritance Models. Genes (Basel). 2018 Apr 16;9(4):215. doi: 10.3390/genes9040215. PMID 29659558
- [Background] Duncan JL, Pierce EA, Laster AM, Daiger SP, Birch DG, Ash JD, Iannaccone A, Flannery JG, Sahel JA, Zack DJ, Zarbin MA; and the Foundation Fighting Blindness Scientific Advisory Board. Inherited Retinal Degenerations: Current Landscape and Knowledge Gaps. Transl Vis Sci Technol. 2018 Jul 18;7(4):6. doi: 10.1167/tvst.7.4.6. eCollection 2018 Jul. No abstract available. PMID 30034950
- [Background] Rodrigues GA, Shalaev E, Karami TK, Cunningham J, Slater NKH, Rivers HM. Pharmaceutical Development of AAV-Based Gene Therapy Products for the Eye. Pharm Res. 2018 Dec 27;36(2):29. doi: 10.1007/s11095-018-2554-7. PMID 30591984
- [Background] Lipinski DM, Thake M, MacLaren RE. Clinical applications of retinal gene therapy. Prog Retin Eye Res. 2013 Jan;32:22-47. doi: 10.1016/j.preteyeres.2012.09.001. Epub 2012 Sep 17. PMID 22995954
- [Background] Verbakel SK, van Huet RAC, Boon CJF, den Hollander AI, Collin RWJ, Klaver CCW, Hoyng CB, Roepman R, Klevering BJ. Non-syndromic retinitis pigmentosa. Prog Retin Eye Res. 2018 Sep;66:157-186. doi: 10.1016/j.preteyeres.2018.03.005. Epub 2018 Mar 27. PMID 29597005
- [Background] Nauta AJ, Fibbe WE. Immunomodulatory properties of mesenchymal stromal cells. Blood. 2007 Nov 15;110(10):3499-506. doi: 10.1182/blood-2007-02-069716. Epub 2007 Jul 30. PMID 17664353
- [Background] Salehi H, Amirpour N, Razavi S, Esfandiari E, Zavar R. Overview of retinal differentiation potential of mesenchymal stem cells: A promising approach for retinal cell therapy. Ann Anat. 2017 Mar;210:52-63. doi: 10.1016/j.aanat.2016.11.010. Epub 2016 Dec 13. PMID 27986614
- [Background] Holan V, Hermankova B, Krulova M, Zajicova A. Cytokine interplay among the diseased retina, inflammatory cells and mesenchymal stem cells - a clue to stem cell-based therapy. World J Stem Cells. 2019 Nov 26;11(11):957-967. doi: 10.4252/wjsc.v11.i11.957. PMID 31768222
- [Background] Tuekprakhon A, Sangkitporn S, Trinavarat A, Pawestri AR, Vamvanij V, Ruangchainikom M, Luksanapruksa P, Pongpaksupasin P, Khorchai A, Dambua A, Boonchu P, Yodtup C, Uiprasertkul M, Sangkitporn S, Atchaneeyasakul LO. Intravitreal autologous mesenchymal stem cell transplantation: a non-randomized phase I clinical trial in patients with retinitis pigmentosa. Stem Cell Res Ther. 2021 Jan 9;12(1):52. doi: 10.1186/s13287-020-02122-7. PMID 33422139
- [Background] He L, Chen Y, Ke Z, Pang M, Yang B, Feng F, Wu Z, Liu C, Liu B, Zheng X, Wu T, Shu T. Exosomes derived from miRNA-210 overexpressing bone marrow mesenchymal stem cells protect lipopolysaccharide induced chondrocytes injury via the NF-kappaB pathway. Gene. 2020 Aug 15;751:144764. doi: 10.1016/j.gene.2020.144764. Epub 2020 May 16. PMID 32428694
- [Background] Keshtkar S, Azarpira N, Ghahremani MH. Mesenchymal stem cell-derived extracellular vesicles: novel frontiers in regenerative medicine. Stem Cell Res Ther. 2018 Mar 9;9(1):63. doi: 10.1186/s13287-018-0791-7. PMID 29523213
- [Background] Vilaca-Faria H, Salgado AJ, Teixeira FG. Mesenchymal Stem Cells-derived Exosomes: A New Possible Therapeutic Strategy for Parkinson's Disease? Cells. 2019 Feb 2;8(2):118. doi: 10.3390/cells8020118. PMID 30717429
- [Background] Zhao T, Sun F, Liu J, Ding T, She J, Mao F, Xu W, Qian H, Yan Y. Emerging Role of Mesenchymal Stem Cell-derived Exosomes in Regenerative Medicine. Curr Stem Cell Res Ther. 2019;14(6):482-494. doi: 10.2174/1574888X14666190228103230. PMID 30819086
- [Background] Frydrychowicz M, Kolecka-Bednarczyk A, Madejczyk M, Yasar S, Dworacki G. Exosomes - structure, biogenesis and biological role in non-small-cell lung cancer. Scand J Immunol. 2015 Jan;81(1):2-10. doi: 10.1111/sji.12247. PMID 25359529
- [Background] Mead B, Ahmed Z, Tomarev S. Mesenchymal Stem Cell-Derived Small Extracellular Vesicles Promote Neuroprotection in a Genetic DBA/2J Mouse Model of Glaucoma. Invest Ophthalmol Vis Sci. 2018 Nov 1;59(13):5473-5480. doi: 10.1167/iovs.18-25310. PMID 30452601
- [Background] Safwat A, Sabry D, Ragiae A, Amer E, Mahmoud RH, Shamardan RM. Adipose mesenchymal stem cells-derived exosomes attenuate retina degeneration of streptozotocin-induced diabetes in rabbits. J Circ Biomark. 2018 Oct 28;7:1849454418807827. doi: 10.1177/1849454418807827. eCollection 2018 Jan-Dec. PMID 30397416
- [Background] Zhang W, Wang Y, Kong Y. Exosomes Derived From Mesenchymal Stem Cells Modulate miR-126 to Ameliorate Hyperglycemia-Induced Retinal Inflammation Via Targeting HMGB1. Invest Ophthalmol Vis Sci. 2019 Jan 2;60(1):294-303. doi: 10.1167/iovs.18-25617. PMID 30657854
- [Background] Ma M, Li B, Zhang M, Zhou L, Yang F, Ma F, Shao H, Li Q, Li X, Zhang X. Therapeutic effects of mesenchymal stem cell-derived exosomes on retinal detachment. Exp Eye Res. 2020 Feb;191:107899. doi: 10.1016/j.exer.2019.107899. Epub 2019 Dec 19. PMID 31866431
- [Background] Moisseiev E, Anderson JD, Oltjen S, Goswami M, Zawadzki RJ, Nolta JA, Park SS. Protective Effect of Intravitreal Administration of Exosomes Derived from Mesenchymal Stem Cells on Retinal Ischemia. Curr Eye Res. 2017 Oct;42(10):1358-1367. doi: 10.1080/02713683.2017.1319491. Epub 2017 Jun 21. PMID 28636406
- [Background] Elbay A, Ercan C, Akbas F, Bulut H, Ozdemir H. Three new circulating microRNAs may be associated with wet age-related macular degeneration. Scand J Clin Lab Invest. 2019 Oct;79(6):388-394. doi: 10.1080/00365513.2019.1637931. Epub 2019 Jul 5. PMID 31277558
- [Background] Bai L, Shao H, Wang H, Zhang Z, Su C, Dong L, Yu B, Chen X, Li X, Zhang X. Effects of Mesenchymal Stem Cell-Derived Exosomes on Experimental Autoimmune Uveitis. Sci Rep. 2017 Jun 28;7(1):4323. doi: 10.1038/s41598-017-04559-y. PMID 28659587
- [Background] Durani P, Leaper D. Povidone-iodine: use in hand disinfection, skin preparation and antiseptic irrigation. Int Wound J. 2008 Jun;5(3):376-87. doi: 10.1111/j.1742-481X.2007.00405.x. PMID 18593388